CLINICAL TRIAL: NCT02744872
Title: Prospektivt Randomiseret Dobbeltblindt Placebo-kontrolleret Studie af, Calciumkanalblokade påbegyndt Inden Operation: Med Henblik på at Forebygge Ciclosporin Induceret Nefropati Efter Lungetransplantation
Brief Title: Copenhagen Acute Renal Complications After Transplantations Study Group
Acronym: CARCATS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Bo Feldt-Rasmussen, Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2008-004771-22
Record Dates: First submitted 2016-03-30; First posted 2016-04-20 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Disorder Related to Lung Transplantation
Keywords: lung transplantation; chronic renal insufficiency
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Felodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Felodipine (Active Comparator): Tablet Felodipin 10 mg x 1 daily
  Interventions: Drug: Felodipine
- Placebo (Placebo Comparator): Identical placebo once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Felodipine — Felodipine 10 mg once daily or identical placebo
  Arms: Felodipine
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Lung transplanted patients experience marked decrease in renal function post transplant mainly due to cyclosporine induced renal changes. Calcium channel blockers may improve renal function in cyclosporine treated transplant recipients through their effects in avoiding cyclosporine-induced renal vasoconstriction and facilitating renal sodium output.

The aim of this study is to examine if calcium channel blockade administered before lung transplantation prevent cyclosporine induced nephropathy.

The design is an intention to treat randomized double blinded single center study. Patients are randomized to two groups, one that received felodipine and one that receives placebo.

Study population is all patients listed for lung transplantation in Denmark in the study period.

Intervention is tablet felodipine titrated to 10 mg, one daily dose in 12 weeks

Primary endpoint is change in renal function as measured by glomerular filtration rate using chromium-51 labeled ethylenediamine tetraacetic acid (51-Cr-EDTA) in the felodipine treated group compared with the placebo group.

DETAILED DESCRIPTION:
Lung transplanted patients experience marked decrease in renal function post transplant mainly due to cyclosporine induced renal changes.

Calcium channel blockers exert renal effects consisting mainly of renal vasodilation and facilitation of renal excretion of sodium through a direct action on renal tubules. Calcium channel blockers improve renal function in cyclosporine treated transplant recipients through their effects in avoiding cyclosporine-induced renal vasoconstriction and facilitating renal sodium output.

Studies in both animal models and humans have demonstrated that calcium channel blockers maintain or reduce renal vascular resistance and preserve or enhance renal blood flow and glomerular filtration rate (GFR).

The aim of this study is to examine if calcium channel blockade administered before lung transplantation prevent cyclosporine induced nephropathy.

The design is an intention to treat randomized double blinded single center study. Patients are randomized to two groups, one that received felodipine and one that receives placebo.

Study population is all patients listed for lung transplantation in Denmark in the study period.

Sample size calculation estimated that 32 patients are needed, 16 patients in each group, with an estimated dropout incidence of 5 patients in each group. This will be able to detect an estimated 50% reduction in the decrease in measured GFR from 40 ml/min in the placebo group to 20 ml/min in treatment group, 80% power and a two-sided t-test, 5 % significance level.

Intervention is tablet Felodipine titrated to 10 mg, one daily dose in 12 weeks

Renal function is determined by 51-Cr-EDTA clearance measurement at times 0 before transplantation and after 1, 3 and 12 weeks.

Primary endpoint is change in renal function as measured by 51-Cr-EDTA clearance in the felodipine treated group compared with the placebo group.

Safety is monitored and adverse events are usually mild headache, tachycardia, leg edema, angina pectoris and hypotension.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are undergoing lung transplantation in Denmark

Exclusion Criteria:

* Fertile women not using contraceptives
* Patients allergic to calcium antagonists
* Patients receiving treatment with Calcium antagonist 14 days prior to transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-09; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in glomerular filtration rate | week 1, 2, 3 and 12
  glomerular filtration rate using chromium-51 labeled ethylenediamine tetraacetic acid (51-Cr-EDTA) at week 1, 2, 3 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Bo Feldt-Rasmussen, Principal Investigator — Professor
Locations (1):
- Department of Nephrology P, Copenhagen University Hospital, Rigshospitalet, Copenhagen Ø, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided